CLINICAL TRIAL: NCT06894498
Title: Five PLus Year EffIcacy of Endoscopic Sleeve Gastroplasty (ESG) for Sustained WeigHT Loss
Acronym: LIGHT
Status: Not yet recruiting | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: E1754
Record Dates: First submitted 2025-03-19; First posted 2025-03-25 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Obesity and Obesity-related Medical Conditions; Weight Loss
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No Intervention: Observational Cohort — No Intervention, Observational Cohort

SUMMARY:
The objective of this study is to assess the long term weight loss and weight loss journey of patients who received an Endoscopic Sleeve Gastroplasty (ESG) 5 or more years prior to enrollment.

DETAILED DESCRIPTION:
Includes retrospective data collection and one prospective visit

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 18 years of age at the time of the ESG procedure
* Subject with a BMI between 30 kg/m2 and 50 kg/m2, inclusive, at the time of the primary ESG procedure using Overstitch Endoscopic Suturing System
* Subject completed follow-up 1-year from the ESG procedure for weight loss management
* Subject completed or is eligible for follow-up 5-years from the ESG procedure for weight loss management (visit can be collected either retrospectively or prospectively)
* Subject has returned for a minimum of one annual follow-up at the treating site for weight loss management annually between two and four years from the procedure.
* Subject is willing to complete one prospective visit (5 year or 5+ year, as appropriate)
* Subject is able to read, understand, and sign a written Informed Consent Form to participate in the study

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be selected from weight loss or bariatric centers
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects that maintain clinically significant weightloss at five-year visit | TBWL assessed at five-years post ESG
  Mean % Total Body Weight Loss (TBWL) at 5-year visit.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (2):
  - Endeavor Health Evanston Hospital, Evanston, Illinois
  - The University of Texas Health Science Center at Houston, Bellaire, Texas
- CHU de Strasbourg, IHU-Strasbourg, Strasbourg, France
- Mohak hi-tech Specialty Hospital, Indore, Madhya Pradesh, India
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Italy
- Spire Southampton, Southampton, Hampshire, United Kingdom